CLINICAL TRIAL: NCT06790914
Title: Investigation on the Status Quo of Hyperalgesia in Patients After Thoracoscopic Operation and Study on the Effect of Intraoperative Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024KY115
Record Dates: First submitted 2024-11-26; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-07

CONDITIONS: Thoracoscopic Surgery; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flurbiprofen axidate combined with noise-cancelling headphones music (Experimental): 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline 50ml at 60 drops /min; After general anesthesia induction, noise-cancelling headphones (Sony WH-1000XM3) were fully covered with both ears, and MP3 (GoGear, Philips) was connected to play music continuously until the headphones were removed after the operation.
  Interventions: Behavioral: Flurbiprofen axidate combined with noise-cancelling headphones music
- flurbiprofen axidate combined with noise-cancelling earphone (Experimental): 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline 50ml at 60 drops /min; After induction of general anesthesia, noise-cancelling headphones (Sony WH-1000XM3) were applied to cover both ears completely until the headphones were removed at the end of the procedure.
  Interventions: Behavioral: Flurbiprofen axidate combined with noise-cancelling headphones
- Flurbiprofen exate on a drip (Placebo Comparator): 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline at 60 drops /min.
  Interventions: Other: Flurbiprofen exate on a drip

INTERVENTIONS:
Behavioral: Flurbiprofen axidate combined with noise-cancelling headphones music — 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline 50ml at 60 drops /min; After general anesthesia induction, noise-cancelling headphones (Sony WH-1000XM3) were fully covered with both ears, and MP3 (GoGear, Philips) was connected to play music continuously until the headphones were removed after the operation.
  Arms: Flurbiprofen axidate combined with noise-cancelling headphones music
Behavioral: Flurbiprofen axidate combined with noise-cancelling headphones — 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline 50ml at 60 drops /min; After induction of general anesthesia, noise-cancelling headphones (Sony WH-1000XM3) were applied to cover both ears completely until the headphones were removed at the end of the procedure.
  Arms: flurbiprofen axidate combined with noise-cancelling earphone
Other: Flurbiprofen exate on a drip — 30min before induction of general anesthesia, flurbiprofen axidate 50mg+ normal saline at 60 drops /min.
  Arms: Flurbiprofen exate on a drip

SUMMARY:
To explore the status quo and influencing factors of hyperpain in patients after thoracoscopic surgery, and to explore the effect of earphone sound isolation during combined operation of flurbiprofen axidate and binaural beat music played by earphone during combined operation on the intervention of hyperpain after thoracoscopic surgery.

DETAILED DESCRIPTION:
In this study, patients undergoing thoracoscopy radical lung cancer surgery in Union Hospital Affiliated to Fujian Medical University were selected for A randomized controlled trial. Patients were selected according to the inclusion and exclusion criteria, and the patients were randomly divided into group A of flurbiprofen axidate combined with noise-canceling headset music test, group B of flurbiprofen axidate combined with noise-canceling headset test, and the control group for intraoperative intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected by the same group of surgeons to perform thoracoscopic three-hole radical resection of lung cancer
* Patients ≥18 years old, able to communicate effectively and cooperate with the completion of clinical trials
* ASA grade I-III
* Normal hearing; Patients who have not participated in other trials in the last two months

Exclusion Criteria:

* Previous history of thoracic surgery
* History of chronic pain and any intake of analgesics 48 hours before surgery; ● Have a history of mental illness, or have taken psychiatric drugs or received psychological treatment in the past six months
* Deformity of the auricle, inability to wear headphones, and failure to cooperate with this study for any reason
* suffering from concurrent severe organ system diseases and hearing impairment
* Incomplete data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-17 (Actual); Primary Completion 2025-03-17 (Estimated); Study Completion 2025-03-17 (Estimated)

PRIMARY OUTCOMES:
The mechanical pain threshold of the medial forearm of the healthy side and the incision area | The first day before surgery, the first day after surgery, and the second day after surgery
  Von Frey cilia were used to measure the pain threshold of the patients. There were 20 kinds of Von Frey cilia intensity, and the corresponding mechanical pain threshold ranges from 0.008 to 300g. Hyperalgesia occurs when values around the incision and/or in the non-dominant forearm are reduced after surgery compared to before surgery.

SECONDARY OUTCOMES:
Numerical Rating Scale（NRS） | The first day before surgery, the first day after surgery, and the second day after surgery
  NRS is a number from 0 to 10 used instead of words to indicate the severity of pain. Score 0 was no pain; 1 to 3 are classified as mild pain, tolerable, and sleep is not affected; 4 to 6 are classified as moderate pain, which begins to affect the patient's sleep and requires the use of painkillers; 7 ~ 9 is classified as severe pain, patients with unbearable pain, affect appetite, sleep is seriously disturbed, autonomic nerve is disturbed; 10 is severe pain.
The first time additional analgesics (NRS≥4) are required after surgery | Within one day of surgery
  The first time additional analgesics (NRS≥4) are required after surgery
The effective number of PCA pump compressions within 48 h after surgery | Within two days of surgery
  The effective number of PCA pump compressions within 48 h after surgery
Total intraoperative use of remifentanil, sevoflurane, and vasoactive agents. | Within one day of surgery
  Total intraoperative use of remifentanil, sevoflurane, and vasoactive agents.
The number of adverse reactions (nausea, vomiting, hypotension, etc.) within 48 hours after surgery | Within two days of surgery
  The number of adverse reactions (nausea, vomiting, hypotension, etc.) within 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fujian, Fuzhou, China